CLINICAL TRIAL: NCT03991910
Title: Randomised Controlled Trial Into the Role of Ramipril in Fibrosis Reduction in Rheumatic Heart Disease: The RamiRHeD Trial Protocol
Brief Title: The Effect of Ramipril in Suppressing ST2 Expression in Rheumatic Mitral Stenosis Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ade Meidian Ambari, MD, cardiologist, head of cardiovascular prevention and rehabilitation, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RamiRHeD
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Rheumatic Heart Disease; Mitral Stenosis; Rheumatic Mitral Stenosis; Fibrosis; Heart; ACE Inhibitor
Keywords: Rheumatic Heart Disease; Mitral Stenosis; Rheumatic Mitral Stenosis; Valve Fibrosis; ramipril; ST2
MeSH Terms: conditions — Rheumatic Heart Disease; Mitral Valve Stenosis; Fibrosis | interventions — Control Groups; Ramipril

STUDY DESIGN:
Intervention Model Description: pre post test design with placebo control
Who Masked: Participant, Investigator
Masking Description: study participants do not know whether they become treatment group or control group the investigator does not know which participant in each group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): control patients will be given a placebo
  Interventions: Drug: Placebos
- treatment (Experimental): Ramipril 5 mg treatment group
  Interventions: Drug: Ramipril 5Mg Oral Capsule

INTERVENTIONS:
Drug: Placebos — the control group will be given placebo inside a capsule, so study participant won't be able to know the drug and doses inside the capsule (for masking). Placebo will be given until 5 days prior to Mitral valve replacement surgery.
  Other Names: control group
  Arms: control
Drug: Ramipril 5Mg Oral Capsule — the treatment group will be given each Ramipril 2,5 mg inside a capsule as an initial dose, for 2 weeks. If there is no serious adverse effect in the observation period of 2 weeks, Ramipril 5 mg inside a capsule will be given for the next weeks until 5 days before the mitral valve surgery date. Study participant won't be able to know the drug and doses inside the capsule (for masking)
  Other Names: treatment group
  Arms: treatment

SUMMARY:
Objective propose: to investigate the effect of Ramipril in suppressing ST2 (suppression of tumorigenicity 2) in the cardiac mitral valve in patients with Rheumatic Heart Disease. We hypothesized that we hypothesized that ramipril will improve rheumatic mitral valve fibrosis through the downregulation of ST2.

DETAILED DESCRIPTION:
The efficacy of secondary prevention is limited in the prevention of RHD progression. For this reason, new strategies and therapies are needed to prevent the progression of RHD. Neutralizing inflammatory cytokines or antagonizing their receptor function has been considered as a useful therapeutic strategy to treat autoimmune diseases. In this respect, new therapies targeting ST 2 and their receptors as studied in some autoimmune diseases may promise a new approach for patients with RHD. Angiotensin II induces the upregulation of Transforming growth factor β (TGF-β) and latter the binding of IL-33 to sST2 and not to the natural ligand (ST2L). The binding of IL-33 to sST2 will cause fibrogenesis even more. Thus, ACEI is hypothesized to attenuate this vicious cycle through the inhibition of Angiotensin II and consequently increase Bradykinin that furtherly inhibits fibrosis through the negative regulation of angiotensin II activity in Mitogen Activator Protein Kinase (MAPK) pathways through the suppression of the Ca2+ response and the Na+ transportACE inhibitor were agents with anti-fibrosis effects. The investigators keen to investigate the effect of Ramipril in suppressing ST2 expression as biomarkers of fibrosis in cardiac mitral valve in patients with Rheumatic Heart Disease in the National Cardiac Center Harapan Kita hospital Jakarta Indonesia. This study was designed as a randomized clinical trial. Patients with mitral stenosis valvular dysfunction due to rheumatic process planned for cardiac valve replacement surgery were given Ramipril or placebo for a minimum of 12 weeks (3 months). ST2 expression will be analyzed as the fibrosis biomarker in the mitral valve. This study will be conducted in the Department of Cardiology and Vascular Medicine, University Indonesia, National Cardiac Center Harapan Kita Hospital, Jakarta, Indonesia from June 2019

ELIGIBILITY:
Inclusion Criteria:

* Patients with mitral valve stenosis or a combination
* aged more than 18 years
* undergo cardiac valve replacement operation with or without a tricuspid valve repair,
* patients with systolic blood pressure (SBP) ≥ 100 mmHg and diastolic blood pressure (DBP) ≥ 60 mmHg
* passed in medication phase without side effect minimum 4 weeks until operation schedule

Exclusion Criteria:

1. Patients with congenital heart disease
2. patients with non-mitral valve surgery
3. patients with coronary artery bypass surgery
4. patients who refuse to join this study.
5. adults aged over 65 years or older
6. pregnant women
7. patients with autoimmune disease.
8. Patients with persistent hypotension (systolic blood pressure (BP) < 100 mm Hg)
9. severe aortic stenosis (aortic valve orifice < 0.75 cm2 )
10. chronic renal dysfunction with serum creatinine > 2.5 mg/ dL,
11. known ACEI intolerance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-06-27 (Actual); Primary Completion 2024-08-08 (Estimated); Study Completion 2024-08-08 (Estimated)

PRIMARY OUTCOMES:
ST2 expression in mitral valve tissue and papillary muscle | a year
  expression of ST2 in mitral valve tissue, using immunohistochemistry method

SECONDARY OUTCOMES:
ST2 Plasma concentration | a year
  plasma level of ST2 measured by ELISA
NT-proBNP concentration (pg/ml) | a year
  concentration of NT-proBNP, plasma markers for cardiac dysfunction.
NYHA class | a year
  related symptoms will be graded in class I to IV according to NYHA.
cardiovascular mortality | 1 year
  Study participants will be followed up until 1 year after the surgery for any mortality that is caused by progression of the cardiac disease
All-cause mortality | 1 year
  Study participants will be followed up until 1 year after the surgery for mortality of any cause.
End diastolic dimension | 1 year
  The diameter across a ventricle at the end of diastole, if not else specified then usually referring to the transverse (left-to-right) internal (luminal) distance, excluding thickness of walls, although it can also be measured as the external distance.
End systolic dimension | 1 year
  The diameter across a ventricle at the end of systole, if not else specified then usually referring to the transverse (left-to-right) internal (luminal) distance, excluding thickness of walls, although it can also be measured as the external distance.
Mitral valve area | 1 year
  mitral valve area is the area of mitral valve, measured by the Gorlin formula MVA (cm2) = (CO ÷ DFP) ÷ (38.0 x MPG) where MVA is the mitral valve area, CO is cardiac output, DFP is the diastolic flow period, 38.0 is the constant and MPG is pressure gradient.
Mitral valve gradient | 1 year
  mitralvalve graient is a echocardiographic parameters of the pressure gradient in the mitral valve
Tricuspid maximal velocity (Vmax) | 1 year
  Tricuspid maximal velocity (Vmax) is the echocardiographic parameters of the maximal velocity in tricuspid valve annulus
Tricuspid regurgitation severity | 1 year
  TRicuspid regurgitation severity is classified ad mild, moderate, and severe, according to European Association of Echocardiography measurement year 2010 for Tricuspid Valve regusrgitation severity.
Ejection fraction | 1 year
  echocardiographic parameter to asses ventricular function
TAPSE (tricuspid annular plane systolic excursion) | 1 year
  echocardiography parameter to asses right ventricular function

CONTACTS AND LOCATIONS:
Overall Officials: Ade Meidian Ambari, MD,FIHA, Principal Investigator — Universitas Indonesia, RSPJN harapan kita
Locations (1):
- Ade Meidian Ambari, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wei Q, Liu H, Liu M, Yang C, Yang J, Liu Z, Yang P. Ramipril attenuates left ventricular remodeling by regulating the expression of activin A-follistatin in a rat model of heart failure. Sci Rep. 2016 Sep 19;6:33677. doi: 10.1038/srep33677. PMID 27642098
- [Background] Shi Q, Abusarah J, Baroudi G, Fernandes JC, Fahmi H, Benderdour M. Ramipril attenuates lipid peroxidation and cardiac fibrosis in an experimental model of rheumatoid arthritis. Arthritis Res Ther. 2012 Oct 18;14(5):R223. doi: 10.1186/ar4062. PMID 23079082
- [Background] Ciccone MM, Cortese F, Gesualdo M, Riccardi R, Di Nunzio D, Moncelli M, Iacoviello M, Scicchitano P. A novel cardiac bio-marker: ST2: a review. Molecules. 2013 Dec 11;18(12):15314-28. doi: 10.3390/molecules181215314. PMID 24335613
- [Background] Ambari AM, Setianto B, Santoso A, Radi B, Dwiputra B, Susilowati E, Tulrahmi F, Doevendans PA, Cramer MJ. Angiotensin Converting Enzyme Inhibitors (ACEIs) Decrease the Progression of Cardiac Fibrosis in Rheumatic Heart Disease Through the Inhibition of IL-33/sST2. Front Cardiovasc Med. 2020 Jul 28;7:115. doi: 10.3389/fcvm.2020.00115. eCollection 2020. PMID 32850979
- [Derived] Ambari AM, Setianto B, Santoso A, Radi B, Dwiputra B, Susilowati E, Tulrahmi F, Wind A, Cramer MJM, Doevendans P. Randomised controlled trial into the role of ramipril in fibrosis reduction in rheumatic heart disease: the RamiRHeD trial protocol. BMJ Open. 2021 Sep 13;11(9):e048016. doi: 10.1136/bmjopen-2020-048016. PMID 34518254